CLINICAL TRIAL: NCT07219589
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HM17321 in Healthy Adult Participants
Brief Title: A SAD Study of HM17321 in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: HM-UCN2-101
Record Dates: First submitted 2025-10-16; First posted 2025-10-22 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Obese
Keywords: Obese; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Participants in each cohort will be randomly assigned to receive either HM17321 or placebo. Dose levels will be escalated sequentially in separate cohorts after review of safety data.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be conducted in a double-blind manner. Participants, investigators, and outcome assessors will remain blinded to treatment assignments. Only designated unblinded personnel (e.g., pharmacist or site staff responsible for drug preparation) will have access to treatment allocation information, and they will not be involved in any other study assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HM17321 (Experimental)
  Interventions: Drug: HM17321
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo of HM17321

INTERVENTIONS:
Drug: HM17321 — Participants will receive a single subcutaneous injection of HM17321 at the assigned dose level. HM17321 is provided as a sterile solution in prefilled syringes.
  Arms: HM17321
Drug: Placebo of HM17321 — Participants will receive a single subcutaneous injection of a matching placebo solution in prefilled syringes. The placebo does not contain any active ingredients.
  Arms: Placebo

SUMMARY:
This is a Phase 1 study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of HM17321 after single ascending doses in healthy adult participants.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, single ascending dose study designed to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of HM17321 in healthy adult participants.

The study will enroll approximately 40 healthy adults with a body mass index (BMI) of ≥20 kg/m² and ≤27 kg/m². Participants will be assigned to 1 of 5 cohorts, with each cohort consisting of 8 participants (6 receiving HM17321 and 2 receiving placebo). The total sample size may be adjusted if additional dose cohorts are added and/or existing cohorts are expanded. Participants who discontinue for reasons other than safety may be replaced at the discretion of the Sponsor and Investigator.

All study drugs will be administered by subcutaneous (SC) injection into the abdominal wall.

The study will include a 28-day screening period, a 5-day inpatient stay during which a single SC dose of HM17321 or placebo will be administered, and an outpatient/follow-up period through Day 29. The study duration for each participant will be approximately 8 weeks from screening to the last follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.
* BMI ≥20 kg/m² and ≤27 kg/m².
* Stable body weight (<5% change) in the past 3 months.
* Able and willing to provide written informed consent.
* Male participants must use contraception or remain abstinent from women of childbearing potential.
* Female participants must not be pregnant or breastfeeding and use effective contraception if of childbearing potential.

Exclusion Criteria:

* History of any bariatric procedure.
* Uncontrolled thyroid disease (TSH >6.0 or <0.4 mIU/L).
* Abnormal liver function tests (ALT or AST >2×ULN, or total bilirubin >1.5×ULN) or severe active liver disease.
* Abnormal pancreatic function (amylase or lipase >3×ULN).
* Clinically significant cardiovascular disorders (e.g., myocardial infarction, congestive heart failure, long QT syndrome).
* Abnormal renal function (eGFR <60 mL/min/1.73 m²).
* Positive test for hepatitis B, hepatitis C, or HIV at screening.
* Women who are pregnant, planning to become pregnant, or breastfeeding.
* History of drug or alcohol abuse within defined timeframes (e.g., alcohol >14 standard units/week in past year, or positive drug screen).
* Use of any investigational product within 30 days or 5 half-lives (whichever is longer) prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events Following a Single Subcutaneous Dose of HM17321 | Up to Day 29
  Number and type of treatment-emergent adverse events and changes in vital signs and laboratory tests up to Day 29

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of HM17321 | Up to Day 29
  Maximum observed plasma concentration after single SC dose up to Day 29.
Time to Maximum Plasma Concentration (Tmax) of HM17321 | Up to Day 29
  Time to maximum observed plasma concentration after single SC dose up to Day 29.
Area Under Plasma Concentration-Time Curve (AUC) of HM17321 | Up to Day 29
  AUC from time zero to last measurable concentration after single SC dose up to Day 29.

OTHER OUTCOMES:
Pharmacodynamics of HM17321 | Up to Day 29
  Body weight(kg) measured at each assessment time point following a single SC dose of HM17321.

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No